CLINICAL TRIAL: NCT03039491
Title: Immune Response to Pneumococcal Vaccination in Aging HIV Positive Individuals
Brief Title: Immune Response to Pneumococcal Vaccination in Aging HIV Positive Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MUSC vaccine study
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: HIV Lipodystrophy; Aging
Keywords: pneumococcal vaccination
MeSH Terms: interventions — Pneumococcal Vaccines; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- HIV+ 50-65, CD4>200 PCV/PPV (Experimental): HIV+ individuals , 50-65 years of age with a nadir cluster of differentiation (CD) 4 count >200 to receive PCV13 vaccine followed 8 weeks later by PPV23
  Intervention: 13 valent Pneumococcal conjugate vaccine (PCV13) followed 8 weeks later by 23 valent pneumococcal polysaccharide vaccine
  Interventions: Biological: Pneumococcal polysaccharide vaccine 23 valent; Biological: 13 valent conjugated pneumococcal vaccine
- HIV+ 50-65, CD4<200 PCV/PPV (Experimental): HIV+ individuals , 50-65 years of age with a nadir CD4 count <200 to receive PCV13 vaccine followed 8 weeks later by PPV23
  Intervention: 13 valent Pneumococcal conjugate vaccine (PCV13) followed 8 weeks later by 23 valent pneumococcal polysaccharide vaccine
  Interventions: Biological: Pneumococcal polysaccharide vaccine 23 valent; Biological: 13 valent conjugated pneumococcal vaccine
- HIV+ 50-65, CD4>200 PPV (Experimental): HIV+ individuals , 50-65 years of age with a nadir CD4 count >200 to receive PPV23 only
  Intervention: 23 valent pneumococcal polysaccharide vaccine only
  Interventions: Biological: Pneumococcal polysaccharide vaccine 23 valent
- HIV+ 50-65, CD4<200 PCV (Experimental): HIV+ individuals , 50-65 years of age with a nadir CD4 count <200 to receive PPV23 only
  Intervention: 23 valent pneumococcal polysaccharide vaccine only
  Interventions: Biological: Pneumococcal polysaccharide vaccine 23 valent
- HIV- 50-65, PCV/PPV (Active Comparator): HIV- individuals , 50-65 years of age immunized with PCV13 followed by PPV23
  Intervention: 13 valent Pneumococcal conjugate vaccine (PCV13) followed 8 weeks later by 23 valent pneumococcal polysaccharide vaccine
  Interventions: Biological: Pneumococcal polysaccharide vaccine 23 valent; Biological: 13 valent conjugated pneumococcal vaccine
- HIV- 50-65, PPV (Active Comparator): HIV- individuals, 50-65 years of age immunized with PPV23 only.
  Intervention: 23 valent pneumococcal polysaccharide vaccine only
  Interventions: Biological: Pneumococcal polysaccharide vaccine 23 valent
- HIV+ 21-40, CD4>200 PCV/PPV (Active Comparator): HIV+ individuals , 21-40 years of age with a nadir CD4 count >200 to receive PCV13 vaccine followed 8 weeks later by PPV23
  Intervention: 13 valent Pneumococcal conjugate vaccine (PCV13) followed 8 weeks later by 23 valent pneumococcal polysaccharide vaccine
  Interventions: Biological: Pneumococcal polysaccharide vaccine 23 valent; Biological: 13 valent conjugated pneumococcal vaccine
- HIV+ 21-40, CD4<200 PCV/PPV (Active Comparator): HIV+ individuals , 21-40 years of age with a nadir CD4 count <200 to receive PCV13 vaccine followed 8 weeks later by PPV23
  Intervention: 13 valent Pneumococcal conjugate vaccine (PCV13) followed 8 weeks later by 23 valent pneumococcal polysaccharide vaccine
  Interventions: Biological: Pneumococcal polysaccharide vaccine 23 valent; Biological: 13 valent conjugated pneumococcal vaccine

INTERVENTIONS:
Biological: Pneumococcal polysaccharide vaccine 23 valent — This is the pneumococcal vaccine consisting of the capsular polysaccharides of 23 serotypes of Streptococcus pneumoniae
  Other Names: Pneumovax
Biological: 13 valent conjugated pneumococcal vaccine — This is the pneumococcal vaccine consisting of the capsular polysaccharides of 13 serotypes of Streptococcus pneumoniae conjugated to non-toxic diphtheria carrier protein 197
  Other Names: Prevnar 13
  Arms: HIV+ 21-40, CD4<200 PCV/PPV; HIV+ 21-40, CD4>200 PCV/PPV; HIV+ 50-65, CD4<200 PCV/PPV; HIV+ 50-65, CD4>200 PCV/PPV; HIV- 50-65, PCV/PPV

SUMMARY:
The investigators hypothesized that pneumococcal vaccination with either the 23-valent pneumococcal polysaccharide vaccine PPV-23 (Pneumovax-23) alone or the 13-valent pneumococcal conjugate vaccine PCV-13 (Prevnar-13) followed by PPV-23 results in a similar antibody levels/functional antibody activity and induce similar pneumococcal polysaccharide (PPS)-specific B cell response in HIV positive individuals > 50 years of age, HIV positive individuals 21-40 years of age as compared to HIV negative > 50 years of age. The investigators immunized the study groups HIV+ persons >50, HIV+ persons 21-40 and controls (HIV negative) with PCV 13 followed by PPV23 and HIV>50 with PPV alone and examined immune responses to polysaccharide (PPS) 23 (F),14, 3, 7 (F) and 19 (A) using polysaccharide specific ELISA and opsonophagocytic assays (OPA). Pre- and post-immunization peripheral blood samples were obtained. Extensive B cell phenotype analysis using fluorescent antibodies was used to characterize PPS-labeled B cells. Specific phenotypes were correlated with antibody levels and OPA and compared to populations immunized with PPV

DETAILED DESCRIPTION:
The purpose of this study is to learn more about how older people with HIV respond to the pneumococcal or pneumonia vaccine. Pneumonia occurs very frequently in in older persons AND in persons who are infected with HIV. Therefore, it is common practice to vaccinate against pneumonia in these patient populations. Because older patients with HIV fit both of these categories, it is believed that they are at an increased risk of pneumonia.

There are two types of pneumonia vaccines available for adults approved by the Federal Drug Administration (FDA). One is called the pneumococcal polysaccharide vaccine (PPV23) and protects against 23 different strains of the pneumonia bacteria. The other type of vaccine called the pneumococcal conjugate vaccine (PCV13) protects against different strains of the pneumonia bacteria.

Until 2012, it was recommended that all HIV-positive adults receive PPV23 when diagnosed with HIV and again 5 years later. More recently, the guidelines have changed to all HIV-positive adults are to receive PCV13, followed later with PPV23. At this point in time, it is not clear which regimen works better in aging HIV positive adults. Investigators are doing this study to compare the effectiveness of each vaccine regimen in aging HIV positive adults compared to healthy adults. Although several studies show short-term efficacy or increased antibody response in HIV+ persons with this vaccine, others do not, in either HIV+ population or in elderly. Large efficacy trials necessary to establish clinical superiority of PCV compared to PPV will likely not be conducted, particularly in the aging HIV+ population. It is therefore essential to define immune responses to conjugated and free-polysaccharide preparations by examining traditional antibody and functional levels as well as B cell subsets, critically affected by aging and HIV. Will either PCV or PPV elicit an immune response compatible with protection in this population? Based on persistent B cell perturbations in HAART-treated persons, it is hypothesized that immunization of aging HIV+ persons with PPV23 will be as effective as a PCV13 containing regimen on a quantitative, qualitative, B and T cell level and that the magnitude of this response will be related to the degree of chronic inflammation. The proposed studies are highly significant as they will define the B and T cell responses to a TI-2 and T-cell dependent form of pneumococcal vaccine in the aging HIV+ population. These data will provide the necessary basis for development of a rational vaccination approach, including the potential use of novel adjuvant. In this study the investigators will:

1. Test the hypothesis that vaccination with either PPV alone (TI-2) or a PCV containing regimen (TD) results in similar antibody levels/functional activity, that are determined by levels of chronic inflammation in aging HIV+. The investigators will immunize the study group HIV+ persons 50-65 and controls (HIV+21-40 and HIV- 50-65 years) with PCV13 followed by PPV23 and HIV+ 50-65 and HIV- 50-65 with PPV alone. The investigators will examine immune responses to pneumococcal polysaccharides (PPS) 23 (F), 14, 3, 7 (F) and 19 (A) on a quantitative and qualitative level using ELISA and opsonophagocytic assays (OPA) and correlate the response to the degree of inflammation measured in each participant.
2. To test the hypothesis that the levels of antigen specific B cells identified with PPS will be comparable between the PPV and PCV vaccine recipients. Pre- and post-immunization peripheral blood samples will be obtained. Extensive phenotype analysis using antibodies against cluster of differentiation (CD)19, 20, 21, 27, 38, 40, immunoglobulin M (IgM) , B-cell activating factor (BAFF), trans-membrane activator and calcium modulator and cyclophilin ligand interactor (TACI), and B-cell maturation antigen (BCMA) markers will be used to characterize PPS-labeled B cells. Specific phenotypes will be correlated with antibody levels, OPA and inflammatory markers and compared to the control populations immunized with PPV.

ELIGIBILITY:
Inclusion Criteria:HIV+ 21-40 years of age HIV+ 50-65 years of age HIV- 50-65 years of age

-

Exclusion Criteria:

* Previous immunization with pneumococcal vaccine less than 5 years ago
* pregnancy and absence of contraceptive practice in women of childbearing age and breast feeding
* known anaphylaxis, hypersensitivity to the pneumonia vaccine
* those who received blood products or gammaglobulin in last 3 months
* inability to comprehend or sihn informed consent
* Medications known to affect immune function (chemotherapy, an angiotensin-converting-enzyme (ACE) inhibitors, corticosteroids, anti-TNFalpha agents)
* previous disease/present illness that may affect response to vaccination: previous pneumococcal disease, removal of spleen, auto-immune disease, end stage renal disease (ESRD) or end stage liver disease, cancer)
* significant (3x upper limit of normal) in complete blood count (CBC), chemistries, immunoglobulin levels

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 160 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Antibody response | Change in ug/mL from day 0 to 30 days after receipt of PPV23
  Measure antibody response by ELISA (ug/mL)
opsonophagocytic antibody activity | Change in opsonophagocytic titer from day 0 to 30 days after receipt of PPV23
  opsonophagocytic antibody response measured by opsonophagocytic assay (OPA)

SECONDARY OUTCOMES:
PPS-specific B cell phenotype | Change from day 0 to day 7 post-vaccination
  Measure: B cell phenotype of PPS-specific B cells expressing CD27+IgM+: flowcytometry (%)
PPS-specific B cell phenotype | Change from day 56 to day 63 post-vaccination
  Measure: B cell phenotype of PPS-specific B cells expressing CD27+IgM+: flowcytometry (%)
Expression of TACI on PPS-specific B cells | change from day 0 to day 7
  Measure:Flow cytometry: percentage of PPS-specific B cells expressing TACI on their surface (%)
Expression of TACI on PPS-specific B cells | change from day 56 to day 63
  Measure:Flow cytometry: percentage of PPS-specific B cells expressing TACI on their surface (%)
Expression of BAFFR on PPS-specific B cells | change from day 0 to day 7
  Measure:Flow cytometry: percentage of PPS-specific B cells expressing BAFFR on their surface (%)
Expression of BAFFR on PPS-specific B cells | change from day 56 to day 63
  Measure:Flow cytometry: percentage of PPS-specific B cells expressing BAFFR on their surface (%)
Expression of BCMA on PPS-specific B cells | change from day 0 to day 7
  Measure:Flow cytometry: percentage of PPS-specific B cells expressing BAFFR on their surface (%)
Expression of BCMA on PPS-specific B cells | change from day 7 to day 63
  Measure:Flow cytometry: percentage of PPS-specific B cells expressing BAFFR on their surface (%)
Expression of CD40 on PPS-specific B cells | change from day 0 to day 7
  Measure:Flow cytometry: percentage of PPS-specific B cells expressing CD40 on their surface (%)
Expression of CD40 on PPS-specific B cells | change from day 56 to day 63
  Measure:Flow cytometry: percentage of PPS-specific B cells expressing CD40 on their surface (%)
Expression of cluster of differentiation 21 (CD21) on PPS-specific B cells | change from day 0 to day 7
  Measure:Flow cytometry: percentage of PPS-specific B cells expressing CD21 on their surface (%)
Expression of CD21 on PPS-specific B cells | change from day 56 to day 63
  Measure:Flow cytometry: percentage of PPS-specific B cells expressing CD21 on their surface (%)
Serum interleukin-6 (IL-6) | Day 0
  Measure serum levels IL-6
Serum BAFF | Day 0
  Measure serum levels BAFF
Serum APRIL | Day 0
  Measure serum levels APRIL
Serum IL-10 | Day 0
  Measure serum levels IL-10
Serum IL-1(RA) | Day 0
  Measure serum levels IL-1RA
Serum IL-1(B) | Day 0
  Measure serum levels IL-1B
Serum IL-8 | Day 0
  Measure serum levels IL-8
Serum TNFalpha | Day 0
  Measure serum levels TNFalpha

CONTACTS AND LOCATIONS:
Overall Officials: Maria A. Julia Westerink, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be made available once analysis is completed through publications in peer reviewed journals.

REFERENCES:
- [Background] Crum-Cianflone NF, Huppler Hullsiek K, Roediger M, Ganesan A, Patel S, Landrum ML, Weintrob A, Agan BK, Medina S, Rahkola J, Hale BR, Janoff EN; Infectious Disease Clinical Research Program HIV Working Group. A randomized clinical trial comparing revaccination with pneumococcal conjugate vaccine to polysaccharide vaccine among HIV-infected adults. J Infect Dis. 2010 Oct 1;202(7):1114-25. doi: 10.1086/656147. PMID 20795819
- [Background] de Roux A, Schmole-Thoma B, Siber GR, Hackell JG, Kuhnke A, Ahlers N, Baker SA, Razmpour A, Emini EA, Fernsten PD, Gruber WC, Lockhart S, Burkhardt O, Welte T, Lode HM. Comparison of pneumococcal conjugate polysaccharide and free polysaccharide vaccines in elderly adults: conjugate vaccine elicits improved antibacterial immune responses and immunological memory. Clin Infect Dis. 2008 Apr 1;46(7):1015-23. doi: 10.1086/529142. PMID 18444818
- [Background] French N, Gordon SB, Mwalukomo T, White SA, Mwafulirwa G, Longwe H, Mwaiponya M, Zijlstra EE, Molyneux ME, Gilks CF. A trial of a 7-valent pneumococcal conjugate vaccine in HIV-infected adults. N Engl J Med. 2010 Mar 4;362(9):812-22. doi: 10.1056/NEJMoa0903029. PMID 20200385
- [Background] Baxendale HE, Keating SM, Johnson M, Southern J, Miller E, Goldblatt D. The early kinetics of circulating pneumococcal-specific memory B cells following pneumococcal conjugate and plain polysaccharide vaccines in the elderly. Vaccine. 2010 Jul 5;28(30):4763-70. doi: 10.1016/j.vaccine.2010.04.103. Epub 2010 May 14. PMID 20471437
- [Background] Penaranda M, Payeras A, Cambra A, Mila J, Riera M; Majorcan Pneumococcal Study Group. Conjugate and polysaccharide pneumococcal vaccines do not improve initial response of the polysaccharide vaccine in HIV-infected adults. AIDS. 2010 May 15;24(8):1226-8. doi: 10.1097/QAD.0b013e3283389de5. PMID 20299956
- [Background] Khaskhely N, Mosakowski J, Thompson RS, Khuder S, Smithson SL, Westerink MA. Phenotypic analysis of pneumococcal polysaccharide-specific B cells. J Immunol. 2012 Mar 1;188(5):2455-63. doi: 10.4049/jimmunol.1102809. Epub 2012 Jan 23. PMID 22271652
- [Derived] Happe M, Samuvel DJ, Ohtola JA, Korte JE, Westerink MAJ. Race-related differences in functional antibody response to pneumococcal vaccination in HIV-infected individuals. Vaccine. 2019 Mar 14;37(12):1622-1629. doi: 10.1016/j.vaccine.2019.01.084. Epub 2019 Feb 21. PMID 30797636